CLINICAL TRIAL: NCT01876797
Title: A Single Dose, Open-label, One Sequence, 2-period, Crossover Study to Characterize the Pharmacokinetics and Pharmacodynamics of Ticagrelor and Prasugrel in Healthy Male Adult Subjects
Brief Title: PKPD Study of Ticagrelor and Prasugrel in Healthy Korean Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hyeong-Seok Lim, Assistant Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Hyeong-Seok Lim
Record Dates: First submitted 2013-06-10; First posted 2013-06-13 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
MeSH Terms: interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ticagrelor-prasugrel (Other): in period 1, 180 mg of ticagrelor will be administrated at a single oral dose. in period 2, 60 mg of prasugrel will be administrated at a single oral dose.
  Interventions: Drug: ticagrelor/prasugrel

INTERVENTIONS:
Drug: ticagrelor/prasugrel
  Other Names: ticagrelor :2 tablets of Brilinta® 90 mg; prasugrel : 6 tablets of Effient® 10 mg

SUMMARY:
This study is to characterize the pharmacokinetic and pharmacodynamics of ticagrelor and prasugrel in healthy Korean male subjects.

The study is open label, one sequence, crossover design. In period 1, a single oral dose of 180 mg ticagrelor will be administrated. After at least 7 days washout period, in period 2, a single oral dose of 60 mg prasugrel will be administrated.

After dosing each period, blood sampling for PK and PD assessment will be conducted.

1. Blood Sampling Times

   1. PK :predose,10 min,15 min,25 min, 0.5,1,1.5,2,2.5,4,6,8,12 and 24h post-dose
   2. PD :predose,15 min,0.5,1,2,4,6,8,12 and 24h post-dose
2. Bioanalysis

   1. plasma Ticagrelor
   2. plasma AR-C124910XX (active metabolite of ticagrelor)
   3. plasma R-95913 (inactive metabolite of prasugrel)
   4. plasma R-13727 (active metabolite of prasugrel)
3. Platelet Aggregation Test using turbidometric Method Maximal Platelet Aggregation(MPA)
4. PK-PD Modeling analysis

ELIGIBILITY:
Inclusion Criteria:

1. male aged 19 - 45 years at screening visit
2. body weight at least 60 kg at screening visit
3. body mass index 18 - 30 kg/m2
4. SBP 90 - 149 mmHg and DBP 60 - 99 mmHg and pulse rate(beat per minute) 45 - 100 at screening visit

Exclusion Criteria:

1. any history of or having any clinically significant abnormalities
2. any gastrointestinal disorder having impact on absorption of study drug
3. any history of hypersensitivity of ticagrelor or prasugrel or compounds related study drugs
4. any history of taking original medicines within 30 days before dosing or history of taking prescribed drug within 14 days before dosing or history of taking OTC drug within 7 days before dosing
5. any history of taking other study drug within 60 days before dosing
6. any history of whole blood transfusion within 60 days before dosing or history of blood elements transfusion or history of heaving been transfused within 30 days before 30 days
7. any history of taking metabolic inducer or inhibitor
8. overuse (caffeine: > 5 units/day , alcohol: > 21 units /week, smoking: > 10 cigarettes/day)
9. positive serology testy(Hbs antigen, HIV, Hepatitis C virus, Syphilis)
10. any abnormality in clinical laboratory tests result or any ECG finding considered to be inadequate by investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
plasma ticagrelor parent,AR-C124910XX,R-95913 and R-13727 | 0,10 min,15 min,25 min,0.5h,1h,1.5h,2h,2.5h,4h,6h,8h,12h and 24h
  4 mL of blood will be drawn per each collection

SECONDARY OUTCOMES:
Maximal Platelet Aggregation(MPA) | 0,15 min,0.5 min, 1h,2h,4h,8h and 24h
  platelet aggregation will be tested using light transmission aggregometry

OTHER OUTCOMES:
adverse event monitoring | up to 1 week
  all adverse event will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Seok Lim, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Jeon HS, Kim MJ, Choi HY, Kim YH, Kim EH, Kim AR, Park HJ, Bae KS, Lim HS. Pharmacokinetics and pharmacodynamics of ticagrelor and prasugrel in healthy male Korean volunteers. Clin Ther. 2015 Mar 1;37(3):563-73. doi: 10.1016/j.clinthera.2015.01.010. Epub 2015 Feb 16. PMID 25697420